CLINICAL TRIAL: NCT05475249
Title: Aesthetic Outcomes of Single Tooth Implant-supported Restorations in the Anterior Maxilla With Either White Zirconia or Fluorescent White Zirconia Abutments: A Randomized Controlled Clinical Study.
Brief Title: Aesthetic Outcomes of Single Tooth Implant-supported Restorations in the Anterior Maxilla With Either White Zirconia or Fluorescent White Zirconia Abutments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Ana Carrillo de Albornoz, Associate Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC14/2017
Record Dates: First submitted 2022-06-27; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Edentulous Alveolar Ridge in the Aesthetic Zone
Keywords: implants AND periodontology AND color OR zirconia AND periimplant mucosa color OR spectrophotometer AND periimplant color

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is designed as double blind, as patient and the clinical examiner (LS) will not have information at any time of which type of abutment is placing, this would be possible due to the identical aspect of both type of abutments. The randomization will be done by the other examiner (AC), that will inform the laboratory.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- white yttria-stabilized zirconia abutment (Placebo Comparator): white yttria-stabilized zirconia abutment (PYRCA; BioHorizons, Birmingham, EEUU) without immersion in fluorescent liquid
  Interventions: Other: Implant placement and prothesis made with different types of abutment
- fluorescence white yttria-stabilized zirconia abutment (Experimental): white yttria-stabilized zirconia abutment (PYRCA; BioHorizons, Birmingham, EEUU) with immersion in fluorescent liquid
  Interventions: Other: Implant placement and prothesis made with different types of abutment

INTERVENTIONS:
Other: Implant placement and prothesis made with different types of abutment — Dental implants (Tapered internal implants; BioHorizons, Birmingham, EEUU) will be placed in healed residual ridges (minimum of 4 months after tooth extraction). After connecting healing abutments, the flaps will be sutured around the abutments for non-submerged healing. An abutment composed of white yttrium oxide stabilized zirconia abutment (PYRCA; BioHorizons, Birmingham, EEUU) previously immersed in fluorescent liquid (Zirkonzahn, South Tirol, Italy) will be placed in the test group, whether in the control group the same abutment will be used but without fluorescent layer. The selected abutment is machined and designed for use with cemented restorations. A single experienced restorative dentist using one dental laboratory carried out all the prosthetic procedures. Single crowns full ceramic will be performed and cemented with RelyX™ Luting Cement.

SUMMARY:
This study aims to answer the question whether the use of a fluorescent layer over white zirconia abutments will improve the aesthetic outcomes of implant borne single-tooth restorations when compared to the use of non-layered white zirconia abutments. The study is designed as a parallel, single-centre and double blind clinical trial. Patients in need of a single tooth implant in the maxilla (from right second premolar to left second premolar, both included) with the presence of adjacent natural teeth will be randomly divided into two treatment groups: using white yttria-stabilized zirconia abutment (PYRCA; BioHorizons, Birmingham, EEUU) with immersion in fluorescent liquid (Zirkonzahn, South Tirol, Italy)(test group) or white yttria-stabilized zirconia abutment (PYRCA; BioHorizons, Birmingham, EEUU) without immersion in fluorescent liquid (control group). 1 and 12 months after crown placement, patients will be recalled and subjected to aesthetic, clinical, radiographic and patient centered outcomes.

DETAILED DESCRIPTION:
Dental implants (Tapered internal implants; BioHorizons, Birmingham, EEUU) will be placed in healed residual ridges (minimum of 4 months after tooth extraction) following the manufacturer's recommendations. After connecting healing abutments, the flaps will be sutured around the abutments for non-submerged healing. A standard postoperative protocol will be followed (antibiotics, anti-inflammatory medication and topical application of 0.12% clorhexidine) and fixed or removable provisional restorations will be provided without immediate occlusal function.

After a 3-months of healing, subjects will be allocated to either test or control group. An abutment composed of white yttrium oxide stabilized zirconia abutment (PYRCA; BioHorizons, Birmingham, EEUU) previously immersed in fluorescent liquid (Zirkonzahn, South Tirol, Italy) will be placed in the test group, whether in the control group the same abutment will be used but without fluorescent layer. The selected abutment is machined and designed for use with cemented restorations.

A single experienced restorative dentist using one dental laboratory will carry out all the prosthetic procedures. Single crowns full ceramic will be performed and cemented with RelyX™ Luting Cement.

The subjects will then be advised to comply with their regular dental hygiene and maintenance protocol and committed to return for one month and one-year examinations in order to register all the outcome variables of the study.

ELIGIBILITY:
Inclusion Criteria:- Systemically and periodontally healthy subjects,18 years of age with good plaque control (less than 25% PlI) or subjects with a healthy periodontium if selected from a periodontal maintenance program.

* The presence of a single tooth gap in the anterior maxilla (from tooth number 1.5-2.5) with the presence of natural adjacent dentition. A minimum 4 months healing was required if the tooth had been recently extracted.
* The presence of ≥ 2 mm of keratinized tissue in the alveolar ridge and enough bone availability to insert a Tapered internal implant (BioHorizons, Birmingham, EEUU) without the need of bone augmentation (minimum of 5.5 mm in width and 9 mm in height).
* The opposing dentition should be stable (without removable appliances) and subjects with bruxism were excluded.

Exclusion Criteria:

* In patients with a history of periodontitis, if periodontitis re-occurred (clinical attachment loss ≥ 2 mm), they will be excluded from the study and receive periodontal therapy.

  * During implant placement, the selected subject will be excluded if implants were not positioned in appropriate prosthetic guided positions. Implants needing any hard tissue augmentation will be excluded before the surgery, however if during the surgery any of this procedure is needed due to unforeseen, the patient will also be excluded from the study "a posteriori".
  * Pregnant women at any time of the study will be excluded.
  * Inadequate vestibular depth to place the Spectrophotometer device

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
The spectrophotometric outcome ΔE is the primary outcome of this study | 1 month after prothesis restoration
  Spectrophotometry (Spectroshade, MTH, Niederhasli, Switzerland) will be used for the color evaluation of the buccal mucosa
The spectrophotometric outcome ΔE is the primary outcome of this study | 1 year after prothesis restoration
  Spectrophotometry (Spectroshade, MTH, Niederhasli, Switzerland) will be used for the color evaluation of the buccal mucosa

SECONDARY OUTCOMES:
Subjective aesthetic outcomes | 1 month after prothesis restoration
  The esthetic index for anterior maxillary implant-supported restorations (CEI) (Juodzbalys et al. 2010) has been selected as visual complex aesthetic index
Subjective aesthetic outcomes | 1 year after prothesis restoration
  The esthetic index for anterior maxillary implant-supported restorations (CEI) (Juodzbalys et al. 2010) has been selected as visual complex aesthetic index
Biological complications | 1 month after prothesis restoration
  Biological complications are considered where there is presence of bleeding on probing (BOP) (peri-implant mucositis) or when BOP is present together with peri-implant bone loss (peri-implantitis)(Lang & Berglund 2011).
Biological Complications | 1 year after prothesis restoration
  Biological complications are considered where there is presence of bleeding on probing (BOP) (peri-implant mucositis) or when BOP is present together with peri-implant bone loss (peri-implantitis)(Lang & Berglund 2011).
Technical complications | 1 month after final prothesis
  Technical complications will be considered as (1) major (requiring replacement of the restoration); such as, implant fracture, abutment tooth fracture, loss of supra-structures, (2) medium; such as abutment fracture, veneer or framework fractures, phonetic complications and (3) minor such as abutment and screw loosening, loss of retention, de-bonding, loss of screw hole sealing or veneer chipping (Lang & Zitzmann 2012).
Technical complications | 1 year after prothesis restoration
  Technical complications will be considered as (1) major (requiring replacement of the restoration); such as, implant fracture, abutment tooth fracture, loss of supra-structures, (2) medium; such as abutment fracture, veneer or framework fractures, phonetic complications and (3) minor such as abutment and screw loosening, loss of retention, de-bonding, loss of screw hole sealing or veneer chipping (Lang & Zitzmann 2012).
Clinical outcomes | Preoperatively
  the mesial and distal adjacent teeth were measured to the nearest 1 mm using a CPC-15 manual periodontal probe (Hu-Friedy, Leinmen, Germany) at 6 six sites per tooth for probing pocket depths (PPD).
Clinical outcomes | Preoperatively
  Full mouth plaque index was recorded.
Clinical outcomes | Preoperatively
  bleeding on probing was recorded.
Clinical outcomes | 1 month after prothesis restoration
  The implant probing depth was measured to the nearest 1 mm using a CPC-15 manual periodontal probe (Hu-Friedy, Leinmen, Germany) at 6 six sites per tooth for probing pocket depths (PPD).
Clinical outcomes | 1 year after prothesis restoration
  The implant probing depth was measured to the nearest 1 mm using a CPC-15 manual periodontal probe (Hu-Friedy, Leinmen, Germany) at 6 six sites per tooth for probing pocket depths (PPD).
Clinical Outcomes | 1 month after final prothesis
  Full mouth plaque index were also be recorded.
Clinical Outcomes | 1 year after final prothesis
  Full mouth plaque index were also be recorded.
Clinical outcomes | 1 month after prothesis restoration
  mucosal recession at the implant (REC) was also recorded
Clinical outcomes | 1 year after prothesis restoration
  mucosal recession at the implant (REC) was also recorded
Clinical outcomes | 1 month after prothesis restoration
  mucosal recession in the adjacent teeth (REC) was also recorded
Clinical outcomes | 1 year after prothesis restoration
  mucosal recession in the adjacent teeth (REC) was also recorded
Radiographic outcomes | 1 year after prothesis restoration
  Standardized intra-oral radiographs were taken using a long-cone paralleling technique and an individualized tooth positioner made of auto-polymerising silicon key (Dentsply Rinn; Elgin, United States). The radiographs were taken immediately after crown placement and at the 12 months follow up. The radiographs were scanned and calibrated using the implant diameter as the fixed reference and the following linear measurements were carried out using image analysis software (NIS-elements software; Nikon, Tokyo, Japan).- Vertical distance (parallel to the implant long axis) from the contact point to the bone crest at mesial and distal sides.
  * Vertical distance from the implant shoulder (placed 1 mm supracrestally) to the most coronal bone in contact with the implant at mesial and distal sites.
  * Horizontal distance from the implant shoulder to the adjacent teeth at mesial and distal sides.
Patient centred outcomes | 1 month after prothesis restoration
  The participating subjects were asked to fill in a written questionnaire for evaluating their satisfaction with regards to the aesthetic appearance, the phonetic ability and their overall satisfaction with the treatment (Pjetursson et al. 2005).
Patient centred outcomes | 1 year after prothesis restoration
  The participating subjects were asked to fill in a written questionnaire for evaluating their satisfaction with regards to the aesthetic appearance, the phonetic ability and their overall satisfaction with the treatment (Pjetursson et al. 2005).

CONTACTS AND LOCATIONS:
Locations (1):
- Leticia, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belser UC, Grutter L, Vailati F, Bornstein MM, Weber HP, Buser D. Outcome evaluation of early placed maxillary anterior single-tooth implants using objective esthetic criteria: a cross-sectional, retrospective study in 45 patients with a 2- to 4-year follow-up using pink and white esthetic scores. J Periodontol. 2009 Jan;80(1):140-51. doi: 10.1902/jop.2009.080435. PMID 19228100
- [Background] Chang M, Odman PA, Wennstrom JL, Andersson B. Esthetic outcome of implant-supported single-tooth replacements assessed by the patient and by prosthodontists. Int J Prosthodont. 1999 Jul-Aug;12(4):335-41. PMID 10635203
- [Background] Dierens M, de Bruecker E, Vandeweghe S, Kisch J, de Bruyn H, Cosyn J. Alterations in soft tissue levels and aesthetics over a 16-22 year period following single implant treatment in periodontally-healthy patients: a retrospective case series. J Clin Periodontol. 2013 Mar;40(3):311-8. doi: 10.1111/jcpe.12049. Epub 2013 Jan 9. PMID 23297745
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Juodzbalys G, Wang HL. Esthetic index for anterior maxillary implant-supported restorations. J Periodontol. 2010 Jan;81(1):34-42. doi: 10.1902/jop.2009.090385. PMID 20059415
- [Background] Lang NP, Zitzmann NU; Working Group 3 of the VIII European Workshop on Periodontology. Clinical research in implant dentistry: evaluation of implant-supported restorations, aesthetic and patient-reported outcomes. J Clin Periodontol. 2012 Feb;39 Suppl 12:133-8. doi: 10.1111/j.1600-051X.2011.01842.x. PMID 22533953
- [Background] Park SE, Da Silva JD, Weber HP, Ishikawa-Nagai S. Optical phenomenon of peri-implant soft tissue. Part I. Spectrophotometric assessment of natural tooth gingiva and peri-implant mucosa. Clin Oral Implants Res. 2007 Oct;18(5):569-74. doi: 10.1111/j.1600-0501.2007.01391.x. Epub 2007 Jul 26. PMID 17655713
- [Background] Pjetursson BE, Zwahlen M, Lang NP. Quality of reporting of clinical studies to assess and compare performance of implant-supported restorations. J Clin Periodontol. 2012 Feb;39 Suppl 12:139-59. doi: 10.1111/j.1600-051X.2011.01828.x. PMID 22533954
- [Background] Pjetursson BE, Karoussis I, Burgin W, Bragger U, Lang NP. Patients' satisfaction following implant therapy. A 10-year prospective cohort study. Clin Oral Implants Res. 2005 Apr;16(2):185-93. doi: 10.1111/j.1600-0501.2004.01094.x. PMID 15777328
- [Background] Sailer I, Zembic A, Jung RE, Siegenthaler D, Holderegger C, Hammerle CH. Randomized controlled clinical trial of customized zirconia and titanium implant abutments for canine and posterior single-tooth implant reconstructions: preliminary results at 1 year of function. Clin Oral Implants Res. 2009 Mar;20(3):219-25. doi: 10.1111/j.1600-0501.2008.01636.x. PMID 19397632
- [Background] Tymstra N, Raghoebar GM, Vissink A, Den Hartog L, Stellingsma K, Meijer HJ. Treatment outcome of two adjacent implant crowns with different implant platform designs in the aesthetic zone: a 1-year randomized clinical trial. J Clin Periodontol. 2011 Jan;38(1):74-85. doi: 10.1111/j.1600-051X.2010.01638.x. Epub 2010 Nov 10. PMID 21062337
- [Background] Zembic A, Bosch A, Jung RE, Hammerle CH, Sailer I. Five-year results of a randomized controlled clinical trial comparing zirconia and titanium abutments supporting single-implant crowns in canine and posterior regions. Clin Oral Implants Res. 2013 Apr;24(4):384-90. doi: 10.1111/clr.12044. Epub 2012 Oct 2. PMID 23025514